CLINICAL TRIAL: NCT03043521
Title: Phase I Study to Investigate Pharmacodynamics of CJ-12420 Compared to Dexlansoprazole With Evening Dosing
Brief Title: Pharmacodynamic Properties of CJ-12420 on Evening Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJ_APA_105
Record Dates: First submitted 2017-01-19; First posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Healthy
MeSH Terms: interventions — Dexlansoprazole; Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CJ-12420 50mg (Experimental): T1=CJ-12420 50mg QD evening (9PM)
  Interventions: Drug: CJ-12420 50mg
- CJ-12420 100mg (Experimental): T2=CJ-12420 100mg QD evening (9PM)
  Interventions: Drug: CJ-12420 100mg
- CJ-12420 200mg (Experimental): T3=CJ-12420 200mg QD evening (9PM)
  Interventions: Drug: CJ-12420 200mg
- Dexlansopazole 60mg (Active Comparator): R=dexlansoprazole 60mg QD evening (9p.m)
  Interventions: Drug: Dexlansoprazole 60 MG

INTERVENTIONS:
Drug: Dexlansoprazole 60 MG
  Other Names: R
  Arms: Dexlansopazole 60mg
Drug: CJ-12420 50mg
  Other Names: T1
  Arms: CJ-12420 50mg
Drug: CJ-12420 100mg
  Other Names: T2
  Arms: CJ-12420 100mg
Drug: CJ-12420 200mg
  Other Names: T3
  Arms: CJ-12420 200mg

SUMMARY:
The purpose of this study is to compare and evaluate impact on pharmacodynamic characteristics of CJ-12420 and dexlansoprazole with evening dosing in healthy male volunteers

DETAILED DESCRIPTION:
Evaluation Criteria:

1. Pharmacokinetic Endpoints Cmax, tmax, AUClast of CJ-12420
2. Pharmacodynamics Endpoints Time pH > 4 Time pH > 6 Integrated acidity Percent inhibition of integrated acidity Percent inhibition time gastric pH ≤ 4 Median pH
3. Safety Assessments Physical examination, ECGs, vital signs (blood pressure, heart rate, body temperature), laboratory test (CBC, Chemistry, UA), and adverse events (AEs)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged ≥20 to ≤45 years
2. Body mass Index (BMI) of 19 to 28kg/m2 ; and a total body weight ≥ 50kg
3. Medically healthy without clinically significant vital signs (blood pressure in sitting position, heart rate)

   * 90 mmHg ≤ Systolic blood pressure (SBP) ≤ 140 mmHg
   * 50 mmHg ≤ Diastolic blood pressure (DBP) ≤ 95 mmHg
   * 45 (beats/min) ≤ Heart rate ≤ 95 (beats/min)
4. Understand restriction during the study and voluntarily consent to participate in the study
5. Consent to use the effective contraceptive methods (using abstinence, spermicide, and condom) and not to donate sperm during the study and until 30 days after completion of study
6. Non-smoker or ex-smoker who stopped smoking for at least one year
7. Negative H. pylori result in urea breath test (UBT)

Exclusion Criteria:

1. History of clinically significant diseases in the digestive, kidney, liver, nervous, hemato-oncologic, endocrine, respiratory, immune, psychiatric, musculoskeletal, or cardiovascular system and other diseases that may harm safety of the subject or may affect the validity of study results, in the judgment of investigator
2. History of allergy or hypersensitivity to any drugs including serious adverse events from treatments such as PPI (omeprazole, rabeprazole, lansoprazole) or P-CAB
3. History surgery that may affect absorption, distribution, metabolism, and elimination of the study drug or in such a medical condition, at the discretion of the principal investigator or sub-investigator
4. History of use of another investigational product within 90 days prior to screening visit
5. Donation of a unit of whole blood within 60 days or blood components or transfusion within 30 days prior to screening visit
6. Having special diet or changes in dietary habits within 30 days prior to screening visit
7. Use of prescription drug within 14 days or over-the-count (OTC) drug including herbal medicine within 7 days prior to screening visit
8. Alcohol > 21 units/week
9. Caffeinated drink intake > 5units/day
10. Positive on urinary drug screening test or urine nicotine test
11. Positive human immunodeficiency virus (HIV), hepatitis B, hepatitis C, or syphilis test
12. Clinically significant abnormal result of liver function (serum ALT, AST or total bilirubin levels ≥ 1.5 times the upper limit of normal (ULN))
13. Inability to tolerate pH catheter insertion
14. History of symptomatic GERD, erosive esophagitis (EE), duodenal ulcer, gastric ulcer, Barrett's esophagus, or Zollinger-Ellison Syndrome
15. Any other conditions which would have made the subject unsuitable for the study in the opinion of the investigator

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male volunteers
Enrollment: 24 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2015-08-12 (Actual); Study Completion 2015-08-12 (Actual)

PRIMARY OUTCOMES:
Time pH > 4 of CJ-12420 | 24 hours pH
  intragastric pH

SECONDARY OUTCOMES:
Cmax of CJ-12420 | up to 20 hours
  maximum measured plasma concentraion
AUClast of CJ-12420 | up to 20 hours
  The area under the plasma concentration versus time curve from time 0 to the last measurable concentration
Cmax of dexlansoprazole | up to 20 hours
  maximum measured plasma concentraion
AUClast of dexlansoprazole | up to 20 hours
  The area under the plasma concentration versus time curve from time 0 to the last measurable concentration
Time pH > 4 of dexlansoprazole | 24 hours pH
  intragastric pH
Median pH > 4 of CJ-12420 | 24 hours pH
  intragastric pH
Median pH > 4 of dexlansoprazole | 24 hours pH
  intragastric pH

CONTACTS AND LOCATIONS:
Overall Officials: Eunji Kim, Study Director — CJ HealthCare Corp.
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No